CLINICAL TRIAL: NCT03302442
Title: Comparison of Oral Molecules Preventing Relapses in Multiple Sclerosis
Acronym: COMP-RMS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0471
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non interventional study — Not applicable - Non interventional Study

SUMMARY:
The aim of this observational study is to compare Dimethyl fumarate (DMF) and Teriflunomide on both clinical and MRI outcomes in patients with relapsing-remitting multiple sclerosis (RRMS) from French Observatory of Multiple Sclerosis (French MS cohort )

ELIGIBILITY:
Inclusion Criteria:

* RRMS Patients with an EDSS score ranging between 0 and 5.5, who initiated either DMF or Teriflunomide before 1/01/2016 and with an available MRI scan and EDSS assessment respectively within 12 and 6 months before treatment initiation Patients who had consent to OFSEP registry Naive patient or treated with prior first line treatment : interferon, glatiramer acetate

Exclusion Criteria:

* Patient with progressive multiple sclerosis
* Patients with prior second line Patient with no MRI or EDSS score within the year before DMF or Teriflunomide initiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RRMS Patients who initiated either DMF or Teriflunomide and with an available MRI scan and EDSS assessment respectively within 12 and 6 months before treatment initiation
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Relapse within first year of treatment | 12 months
  Proportion of patients experimenting at least one relapse within the first year of treatment

SECONDARY OUTCOMES:
Occurrence of clinical event at Two years | 24 months
  Proportion of patients with at least one relapse at two years of treatment
Progression of disability | 12 months and 24 months
  Proportion of patients with a progression of disability defined by any increased of EDSS score compared to baseline
Radiological disease activity | 12 months and 24 months
  Proportion of patients with at least one Gd-enhancing lesion and the proportion of patients with at least one new T2-lesion on MRI scans compared to baseline MRI scan Probablity
Adverse drug reaction | 12 months and 24 months
  Number and description of adverse reaction. Proportion of patients who had stopped treatment due to AR

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No